CLINICAL TRIAL: NCT02921139
Title: Comparing Re-trans-catheter Arterial Chemoembolization Versus Stereotactic Ablative Radiotherapy for Hepatocellular Carcinoma Patients Who Had Incomplete Response After Prior TACE (TASABR Trial): a Randomized Controlled Trial
Brief Title: Comparing Re-TACE Versus SABR for Post-prior-TACE Incompletely Regressed HCC: a Randomized Controlled Trial (TASABR)
Acronym: TASABR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dalin Tzu Chi General Hospital (Other)
Collaborators: Buddhist Tzu Chi General Hospital (Other); Hualien Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A10502001
Record Dates: First submitted 2016-09-29; First posted 2016-10-03 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Hepatocellular Carcinoma(HCC)
Keywords: Hepatocellular Carcinoma; Transcatheter Arterial Chemoembolization (TACE); Stereotactic ablative radiotherapy (SABR)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Stereotactic ablative radiotherapy (SABR)
  Interventions: Radiation: Stereotactic ablative radiotherapy (SABR)
- Arm II (Active Comparator): Re-transcatheter arterial chemoembolization (re-TACE)
  Interventions: Procedure: Re-Transcatheter arterial chemoembolization (re-TACE)

INTERVENTIONS:
Radiation: Stereotactic ablative radiotherapy (SABR) — Patients with HCC after incomplete TACE are randomized to stereotactic ablative radiotherapy (SABR). SABR will be delivered in 5 fractions.The preferred inter-fraction time interval is 48 hours. The entire treatment with 10 days is preferred.
  Other Names: Stereotactic Body Radiation Therapy (SBRT)
  Arms: Arm I
Procedure: Re-Transcatheter arterial chemoembolization (re-TACE) — Patients with HCC after incomplete TACE are randomized to further re-TACE.
  Other Names: Transarterial Chemoembolization
  Arms: Arm II

SUMMARY:
Till now, trans-arterial chemoembolization (TACE) is still one of the common modalities in treating hepatocellular carcinoma patients with unresectable intermediate stage. However, residual viable HCC after TACE is not uncommon, leading to a poor overall survival after TACE alone. Recently, stereotactic ablative radiotherapy (SABR) has been reported to be potentially useful for curatively managing early-stage HCC in retrospective studies. Thus, conducting a randomized clinical trial to test the role of SABR in eradicating post-TACE residual tumors is therefore encouraged. The present phase-III trial intended to compare clinical outcomes between TACE + SABR and TACE + re-TACE for HCC patients with post-prior-TACE residual tumors.

DETAILED DESCRIPTION:
Developing effective treatment modalities is crucial in managing HCC patients with unresectable intermediate stage. Nowadays, many therapies have been used for treating this group of HCC patients, including TACE. However, residual tumors after TACE are not uncommon. In conventional, re-TACE is recommended for managing residual tumors. However, accumulated overall survival is still poor in consecutive TACEs, leading to a low rate of <20% in 5 years.

In this regard, radiotherapy has been proved to be effective in managing HCC patients, especially a novel technique named SABR. When compared with conventional-fractionated radiotherapy, SABR demonstrated better treatment responses with fewer side effects in managing primary or metastatic liver tumors. In the literature, phase I and II trials of TACE plus SABR showed excellent local control rates and promising 1- and 2-year survival rates. However, till now, there is no head-to-head comparison between TACE + SABR and consecutive TACEs.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a) Radiographic enhancing liver lesions with early enhance and delay wash out on triple phase CT or MRI or b) histological confirmation of HCC as determined by the Liver Tumor Board
* Age ≧ 20
* Genders: Both male and female
* Barcelona Clinic Liver Cancer (BCLC) stage A to B
* Child-Pugh A or B
* Unresectable tumors or medically inoperable status or surgery was declined/refused.
* Meets clinical criteria for eligibility for TACE or SABR
* SABR can be applied within 6 weeks of registration
* Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Life expectancy > 12 weeks
* negative pregnancy
* No prior treatment, except for surgical resection and radiofrequency ablation (RFA)
* Lab ：

  1. Hemoglobin ≧ 8.0 g/dL(may be post-transfusion if clinically indicated)
  2. Total bilirubin ≦ 3.0 mg/dL
  3. Aspartate aminotransferase (AST) ≦ 5x institutional upper limit of normal
  4. Alanine transaminase (ALT) ≦ 5x institutional upper limit of normal
  5. Absolute neutrophil count ≧ 1,000 /μl
  6. Platelet count ≧ 20,000/μl (may be post-transfusion if clinically indicated)
  7. Prothrombin time-international normalized ratio ≤ 1.7

Exclusion Criteria:

* Previous TACE ≥ 2 times
* Prior radiotherapy to the upper abdomen
* Prior invasive malignancy other than primary liver malignancy (except non-melanomatous skin cancer) unless disease free for at least 3 years
* metastatic disease
* cardiac ischemia or stroke within last 6 months
* medical or psychosocial condition unsuitable
* History of sorafenib therapy within 21 days prior

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-11; Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
freedom form local progression | Up to 12 months
  The freedom from local progression is defined as no in-field progressive disease. It will be estimated by Kaplan-Meier and Cox regression model adjusting for the competing risks

SECONDARY OUTCOMES:
Overall survival | Up to 24 months
  To estimate the rates of overall survival. It will be estimated by Kaplan-Meier and Cox regression model adjusting for the competing risks
Progression-free survival | Up to 24 months
  To estimate the rates of progression-free survival. It will be estimated by Kaplan-Meier and Cox regression model adjusting for the competing risks
Response rate | Up to 24 months
  To estimate the response rate. It will be estimated by Kaplan-Meier and Cox regression model adjusting for the competing risks
Duration of Response of the treated tumor | Up to 24 months
  The duration of the response is from the time response is achieved until disease progression is detected. It will be estimated by Kaplan-Meier and Cox regression model adjusting for the competing risks
Grade of toxicity | Up to 24 months
  To estimate the rate of acute and late treatment-related toxicity related to specific symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Kai Hung, PhD, Principal Investigator — Chief of Department of Radiation Oncology and Cancer Center, Dalin Tzu Chi Hospital
Locations (1):
- Dalin Tzu Chi Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chang IC, Huang SF, Chen PJ, Chen CL, Chen CL, Wu CC, Tsai CC, Lee PH, Chen MF, Lee CM, Yu HC, Lo GH, Yeh CT, Hong CC, Eng HL, Wang J, Tseng HH, Hsiao CH, Wu HI, Yen TC, Liaw YF. The Hepatitis Viral Status in Patients With Hepatocellular Carcinoma: a Study of 3843 Patients From Taiwan Liver Cancer Network. Medicine (Baltimore). 2016 Apr;95(15):e3284. doi: 10.1097/MD.0000000000003284. PMID 27082566
- [Background] Cheng X, Sun P, Hu QG, Song ZF, Xiong J, Zheng QC. Transarterial (chemo)embolization for curative resection of hepatocellular carcinoma: a systematic review and meta-analyses. J Cancer Res Clin Oncol. 2014 Jul;140(7):1159-70. doi: 10.1007/s00432-014-1677-4. Epub 2014 Apr 22. PMID 24752339
- [Background] Huo YR, Eslick GD. Transcatheter Arterial Chemoembolization Plus Radiotherapy Compared With Chemoembolization Alone for Hepatocellular Carcinoma: A Systematic Review and Meta-analysis. JAMA Oncol. 2015 Sep;1(6):756-65. doi: 10.1001/jamaoncol.2015.2189. PMID 26182200
- [Background] Kang JK, Kim MS, Cho CK, Yang KM, Yoo HJ, Kim JH, Bae SH, Jung DH, Kim KB, Lee DH, Han CJ, Kim J, Park SC, Kim YH. Stereotactic body radiation therapy for inoperable hepatocellular carcinoma as a local salvage treatment after incomplete transarterial chemoembolization. Cancer. 2012 Nov 1;118(21):5424-31. doi: 10.1002/cncr.27533. Epub 2012 May 8. PMID 22570179
- [Background] Takeda A, Sanuki N, Tsurugai Y, Iwabuchi S, Matsunaga K, Ebinuma H, Imajo K, Aoki Y, Saito H, Kunieda E. Phase 2 study of stereotactic body radiotherapy and optional transarterial chemoembolization for solitary hepatocellular carcinoma not amenable to resection and radiofrequency ablation. Cancer. 2016 Jul 1;122(13):2041-9. doi: 10.1002/cncr.30008. Epub 2016 Apr 8. PMID 27062278
- [Background] Wahl DR, Stenmark MH, Tao Y, Pollom EL, Caoili EM, Lawrence TS, Schipper MJ, Feng M. Outcomes After Stereotactic Body Radiotherapy or Radiofrequency Ablation for Hepatocellular Carcinoma. J Clin Oncol. 2016 Feb 10;34(5):452-9. doi: 10.1200/JCO.2015.61.4925. Epub 2015 Nov 30. PMID 26628466
- [Derived] Chen LC, Chiou WY, Lin HY, Lee MS, Lo YC, Huang LW, Chang CM, Hung TH, Lin CW, Tseng KC, Liu DW, Hsu FC, Hung SK. Comparing stereotactic ablative radiotherapy (SABR) versus re-trans-catheter arterial chemoembolization (re-TACE) for hepatocellular carcinoma patients who had incomplete response after initial TACE (TASABR): a randomized controlled trial. BMC Cancer. 2019 Mar 28;19(1):275. doi: 10.1186/s12885-019-5461-3. PMID 30922261